CLINICAL TRIAL: NCT03758391
Title: Comparison of a "Flipped" Classroom Methodology to Traditional Instructional Techniques for Neonatal-perinatal Medicine Fellows: A National Prospective Study
Brief Title: Comparison of Learning in Traditional Versus "Flipped" Classrooms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: American Academy of Pediatrics Section of Neonatal-Perinatal Medicine (Unknown); Organization of Neonatal-Perinatal Medicine Training Program Directors (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-015235
Record Dates: First submitted 2018-11-19; First posted 2018-11-29 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Medical Education
Keywords: Neonatal-Perinatal Medicine; Andragogy; Flipped Classroom

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Didactic Education (No Intervention): Education will be provided to fellows using the traditional didactic approach (lecture-based).
- Flipped Classroom Education (Experimental): Education will be provided to fellows using the flipped classroom approach.
  Interventions: Other: Flipped Classroom education

INTERVENTIONS:
Other: Flipped Classroom education — Fellows will receive GI/Bilirubin education in a flipped classroom format.
  Arms: Flipped Classroom Education

SUMMARY:
This is an educational research study to compare knowledge retention of neonatal-perinatal medicine (NPM) fellowship trainees instructed on a subsection of the American Board of Pediatrics (ABP) NPM Content Outline using traditional didactic lectures (control group) versus a flipped classroom methodology (intervention group). The primary objectives are to assess whether the flipped classroom provides equivalent or superior outcomes for knowledge acquisition and retention compared to traditional lecture-based formats, based upon baseline and serial knowledge assessments (after the educational session, and at 3- and 6- month intervals). The secondary outcomes are learner and educator preference.

DETAILED DESCRIPTION:
Sixty-three ACGME-accredited NPM fellowship training programs in the United States have enrolled to participate in this study. Programs have been randomized to teach a subsection of neonatal physiology using the traditional didactic approach or using the "flipped" classroom methodology.

The ACGME requires that NPM fellowship programs provide formal instruction to teach trainees about key concepts in the care of neonates and infants, and most programs have traditionally utilized didactic presentations to relay this information. These sessions are typically instructor-centered, with little requirement for involvement or engagement on the part of the learner, and are not felt to optimize long-term knowledge acquisition and retention. A newer educational model, the "flipped" classroom, increases the opportunities for learner engagement and requires investment and preparation. Using this educational structure, fellows receive learning materials that need to be reviewed prior to the in-person educational session. The participants will then spend the in-person session actively engaged in applying the knowledge to answer questions, participate in discussions, and solve problems. Adult learning theory supports this active involvement as a way to increase learner engagement, improve recognition of meaning of the material, and improve knowledge acquisition and long-term retention.

Fellowship Program Directors involved in the Organization of Neonatal Training Program Directors (ONTPD) have been contacted about the opportunity to participate in this prospective multi-center study. After enrollment, program directors will complete a brief survey of their program's baseline educational methods and demographics. Fellows will be contacted directly by local site PIs for individual consent to data collection. Fellows will be asked to provide demographic information, assessment of learning style/ practices, time devoted to educational pursuits, and perceptions of current physiology education. The fellows will be asked to complete 4 knowledge assessments (baseline, at the end of the educational block, 3 months, 6 months) in REDCap over the course of 6 months. All data will be de-identified, and individual and programmatic data will be anonymous. The assigned ABP content will be taught within the same 3-month period any time between September 2018 and March 2019 via the assigned method (traditional didactic or flipped classroom). All educational materials will be provided to both arms of the study. Learning objectives will be based on the ABP NPM Content Outline and materials with be authored by experts in neonatal physiology. Materials will undergo rigorous peer-review by an editorial board. Traditional/control fellows will be instructed using the provided educational materials in an instructor-led didactic slide presentation. Intervention group fellows will be required to view the same educational materials in online videos prior to their assigned classroom session. During the "flipped" classroom session, the fellows will work through a series of questions based on the assigned educational materials with a local facilitator using a facilitation guide who has been trained in flipped classroom facilitation. This facilitator guide will present discussion points based upon the pre-learning materials and requires learners to apply acquired knowledge. The facilitator guides are also peer-reviewed for content and quality.

In the present study, only the ABP Content Objectives for NPM on gastroenterology and bilirubin will be included. Educational materials will be reviewed and revised by a 4-member editorial board to ensure accuracy, completeness, and quality. For online viewing, these materials are uploaded on MedEdOnTheGo.com, an online learning management platform. Fellows will be provided with additional reading materials, such as seminal articles or textbook chapters, that will allow them to develop a deep understanding of the topic.

Fellows will be surveyed regarding their learning experiences at 3 different time points; before the educational intervention begins, at the completion of the educational intervention, and 3 months after completion of the intervention. Fellows will complete anonymous surveys in REDCap regarding their learning experiences, class preparation, the quality of teaching, perceived effectiveness of teaching efforts, and preferences for learning. Fellows will also participate in short 15-item multiple choice quizzes to measure knowledge retention. There will be 4 quizzes in total; prior to the intervention (baseline), at the completion of the intervention, 3 months post, and 6 months post-intervention. These quizzes will be proctored and closed book. Fellows in either randomization arm will answer the same questions. The quiz questions will cover the specific content addressed in the educational sessions, be created by the study team, and piloted by attending neonatologists for clarity, accuracy, and relevance.

Data will be tabulated on baseline information for both program level and fellow level with testing to determine if pre-intervention testing data is different between groups (equivalence variance 2-tailed T-tests for continuous data and likert scores, and chi square for categorical data). Knowledge retention curves will be developed by performing T-tests of mean scores for each time point. Post-education surveys for program directors and fellows will be evaluated to assess effect of interventions using equal variance 2-tailed T-tests for continuous data and likert scores.

ELIGIBILITY:
Inclusion Criteria:

* Fellow or educator in an ACGME-accredited Neonatal-Perinatal Medicine Fellowship program in the US.

Exclusion Criteria:

* Not a fellow or educator in an ACGME-accredited Neonatal-Perinatal Medicine Fellowship program in the US.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Knowledge retention | 9 months
  Knowledge retention will be tested using multiple choice examinations.

SECONDARY OUTCOMES:
Learner Preferences | 6 months
  Learner preferences for how to receive education will be assessed through qualitative survey
Educator Preferences | 6 months
  Educator preferences for how to provide education will be assessed through qualitative survey

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States